CLINICAL TRIAL: NCT02878538
Title: An N of One Clinical Trial to Pilot the Feasibility of Using the Iron-Chelator Deferiprone on Mild Cognitive Impairment
Brief Title: A Pilot of the Feasibility of Using the Iron-Chelator Deferiprone on Mild Cognitive Impairment
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study was withdrawn before IRB approval
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: P30AG044271 (NIH); HSC20160395H (Other: University of Texas Health Science Center- San Antonio)
Record Dates: First submitted 2016-08-05; First posted 2016-08-25 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2017-08

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Deferiprone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- deferiprone (Active Comparator): Deferiprone will be administered three times a day (25mg/kg). Total dose per day will depend on participants' body weight for one, three month block.
  Interventions: Drug: Deferiprone
- Placebo Phase (Placebo Comparator): Placebo tablets with inactive substance will be used. Total number of placebo tablets will be equivalent to the active tablets administered depending on participants' body weight for two, three month blocks.
  Interventions: Other: Placebo phase

INTERVENTIONS:
Drug: Deferiprone — Subjects will then begin an experimental No1 design: placebo-deferiprone-placebo. Study drug will be administered in three 3 month blocks. All subjects will receive 30 days of active study drug. The placebo-deferiprone contrast compares placebo to active drug initiation. The deferiprone-placebo contrast tests active drug withdrawal. All will be given placebo in months 1-3, and 6-12. This will allow the investigators to examine active drug exposure on d score up to one year and prospective time to MCI conversion. Dosing: Participants will be treated 25 mg/kg po tid (75mg /kg /d total) The dose will be rounded by the prescriber to the nearest 250 mg (half-tablet).
  Other Names: Ferriprox, ATC Code V03AC02
  Arms: deferiprone
Other: Placebo phase — Placebo tablets with inactive substance will be provided to subjects for two, 3 month blocks during the study.
  Arms: Placebo Phase

SUMMARY:
The investigators propose to conduct a series of N of One (No1) single blinded clinical trials to pilot the feasibility of using the iron-chelator deferiprone on Mild Cognitive Impairment (MCI). Chelation therapy has previously been reported to slow the rate of cognitive decline in Alzheimer's Disease (AD) by 50% in a single human randomized clinical trial.

DETAILED DESCRIPTION:
Iron chelation's mechanism of action (MOA) in Alzheimer's disease (AD) is uncertain. Potential MOA include reversal of aluminum (AL) toxicity, the prevention of a-beta aggregation, β-amyloid disaggregation, and the obstruction of microbacterial and viral parasitism. The latter mechanism involves augmentation of innate immunity, and disruption of microbacterial iron metabolism. Infectious models of AD's pathophysiology have been recently proposed. Iron blocks toll-like receptor (TLR) initiated anti-microbial actions mediated via gamma-interferon (IFN-γ) tumor necrosis factor alpha (TNF-alpha), interleukin-6 (IL-6), and interleukin-10 (IL-10). These biomarkers are of interest because they have also been associated with our novel latent dementia phenotype (i.e., "d" for "dementia") in the Texas Alzheimer's Research and Care Consortium (TARCC). "d" is a continuous measure of dementia severity that can be constructed from any cognitive battery that also includes a measure of Instrumental Activities of Daily Living (IADL). Serum biomarkers might "trigger" dementing processes without participating in their later stages. Thus, the investigators have indications as to who might benefit from iron-chelation and when the intervention might be best applied. This knowledge may help them detect an effect of deferiprone on prospective change in "d" and even on MCI conversion in TARCC NHW (Non Hispanic White) subjects.

ELIGIBILITY:
Inclusion Criteria:

1. MA (Mexican Americans) or NHW TARCC participants with competent informants;
2. TARCC diagnosis of "MCI" (any subtype);
3. Incident MCI or conversion to MCI from control in the two previous TARCC waves;
4. 65-80 yrs of age;
5. Non-institutionalized level of care;
6. Capacity to give informed consent
7. GDS (Geriatric Depression Screen) score (15 item) ≤ 6;
8. TARCC MMSE (Mini-Mental State Examination) ≥ 26 /30;
9. HIS (Hachinski Ischemic Scale) ≤ 05/15;
10. Most recent TARCC dEQ-score = 0 ± 0.25.

Exclusion Criteria:

1. A clinical diagnosis of "Diabetes Mellitus" and current treatment with insulin;
2. A self-reported diagnosis of "Major Depression" (treatment with "antidepressants" not exclusionary);
3. A history of psychosis, including visual hallucinations;
4. History or treatment for Parkinson's, or tremor, or Rapid Eye Movement (REM) behavior disorder;
5. History or treatment for atrial fibrillation;
6. Treatment for cancer in the last 5 years (exc. skin cancers);
7. Major surgery in the last year;
8. History of craniotomy;
9. Serum Ferritin < 500mcg/ml, Hgb < 14g/dl♂ /12g/dl♀,, HCT < 45%♂ /40%♀, recent blood transfusion (last 5 years), FeSO4 supplementation, erythromycin therapy;
10. ANC (absolute neutrophil count) < 500 cells/µL, platelet count < 150 × 106 /ml;
11. Treatment with anti-convulsants, mood stabilizers, neuroleptics, opiates, muscle relaxants, systemic steroids, or AD-indicated agents.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Efficacy of deferiprone therapy on "d" scores in Mild Cognitive Impairment (MCI) | 12 months
  Using N of 1 trial design in small number of MCI cases to compare within subject response to placebo and deferiprone in a A1-A-A1 design

SECONDARY OUTCOMES:
Explore deferiprone's longitudinal effect on "d" and dementia conversion | 12 months
  We want to survey the effect of deferiprone on "d" to see If serum biomarkers trigger dementing processes in non Hispanic whites and if deferiprone exposure in MCI may terminate progression and conversion to dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Donald R Royall, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio; Dean Kellogg, MD, PHD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Becerril-Ortega J, Bordji K, Freret T, Rush T, Buisson A. Iron overload accelerates neuronal amyloid-beta production and cognitive impairment in transgenic mice model of Alzheimer's disease. Neurobiol Aging. 2014 Oct;35(10):2288-301. doi: 10.1016/j.neurobiolaging.2014.04.019. Epub 2014 May 1. PMID 24863668
- [Background] De Chiara G, Marcocci ME, Sgarbanti R, Civitelli L, Ripoli C, Piacentini R, Garaci E, Grassi C, Palamara AT. Infectious agents and neurodegeneration. Mol Neurobiol. 2012 Dec;46(3):614-38. doi: 10.1007/s12035-012-8320-7. Epub 2012 Aug 17. PMID 22899188
- [Background] Fine JM, Renner DB, Forsberg AC, Cameron RA, Galick BT, Le C, Conway PM, Stroebel BM, Frey WH 2nd, Hanson LR. Intranasal deferoxamine engages multiple pathways to decrease memory loss in the APP/PS1 model of amyloid accumulation. Neurosci Lett. 2015 Jan 1;584:362-7. doi: 10.1016/j.neulet.2014.11.013. Epub 2014 Nov 13. PMID 25445365
- [Background] Gavett BE, Vudy V, Jeffrey M, John SE, Gurnani AS, Adams JW. The delta latent dementia phenotype in the uniform data set: Cross-validation and extension. Neuropsychology. 2015 May;29(3):344-52. doi: 10.1037/neu0000128. Epub 2014 Aug 25. PMID 25151112
- [Background] Hughes CP, Berg L, Danziger WL, Coben LA, Martin RL. A new clinical scale for the staging of dementia. Br J Psychiatry. 1982 Jun;140:566-72. doi: 10.1192/bjp.140.6.566. PMID 7104545
- [Background] Nairz M, Schroll A, Sonnweber T, Weiss G. The struggle for iron - a metal at the host-pathogen interface. Cell Microbiol. 2010 Dec;12(12):1691-702. doi: 10.1111/j.1462-5822.2010.01529.x. Epub 2010 Oct 21. PMID 20964797
- [Background] Peters DG, Connor JR, Meadowcroft MD. The relationship between iron dyshomeostasis and amyloidogenesis in Alzheimer's disease: Two sides of the same coin. Neurobiol Dis. 2015 Sep;81:49-65. doi: 10.1016/j.nbd.2015.08.007. Epub 2015 Aug 22. PMID 26303889
- [Background] Royall DR, Palmer RF, Markides KS. Exportation and Validation of Latent Constructs for Dementia Case Finding in a Mexican American Population-based Cohort. J Gerontol B Psychol Sci Soc Sci. 2017 Oct 1;72(6):947-955. doi: 10.1093/geronb/gbw004. PMID 26968639
- [Background] Royall DR, Palmer RF; Texas Alzheimer's Research and Care. Validation of a latent construct for dementia case-finding in Mexican-Americans. J Alzheimers Dis. 2013;37(1):89-97. doi: 10.3233/JAD-130353. PMID 23800829
- [Background] Royall DR, Palmer RF. Ethnicity moderates dementia's biomarkers. J Alzheimers Dis. 2015;43(1):275-87. doi: 10.3233/JAD-140264. PMID 25079802
- [Background] Royall DR, Palmer RF. Thrombopoietin is associated with delta's intercept, and only in Non-Hispanic Whites. Alzheimers Dement (Amst). 2016 Feb 26;3:35-42. doi: 10.1016/j.dadm.2016.02.003. eCollection 2016. PMID 27239547
- [Background] Royall DR, Palmer RF, O'Bryant SE; Texas Alzheimer's Research and Care Consortium. Validation of a latent variable representing the dementing process. J Alzheimers Dis. 2012;30(3):639-49. doi: 10.3233/JAD-2012-120055. PMID 22451315
- [Background] Salkovic-Petrisic M, Knezovic A, Osmanovic-Barilar J, Smailovic U, Trkulja V, Riederer P, Amit T, Mandel S, Youdim MB. Multi-target iron-chelators improve memory loss in a rat model of sporadic Alzheimer's disease. Life Sci. 2015 Sep 1;136:108-19. doi: 10.1016/j.lfs.2015.06.026. Epub 2015 Jul 6. PMID 26159898